CLINICAL TRIAL: NCT00322140
Title: Phase I Study of CDDO in Solid Tumors and Lymphomas
Brief Title: CDDO to Treat Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060151; 06-C-0151; NCT00352040 (obsolete NCT alias)
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08-25

CONDITIONS: Solid Tumors; Lymphoma
Keywords: Metastatic; Triterpenoids; 2-Cyano-3,12-Dioxooleana-1,9(11)Dien-28oic Acid; Dose-Limiting; Pharmacokinetic; Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma; Neoplasm Metastasis | interventions — bardoxolone

INTERVENTIONS:
Drug: CDDO

SUMMARY:
Background:

* CDDO is a novel synthetic triterpenoid which is a potent multifunctional molecule. It induces apoptosis in vitro in malignant cells through both intrinsic and extrinsic pathways, and it controls cellular differentiation, apoptosis, and growth inhibition by serving as a ligand for the transcription factor peroxisome proliferator activator receptor-gamma (PPAR gamma).
* Based on in vitro activity, it holds considerable promise as a novel anti-tumor agent against a wide range of malignancies by concurrently targeting multiple pathways leading to oncogenesis.
* In vivo data demonstrates that the drug is well tolerated in dogs, and has anti-tumor effects, dependent upon dose schedule.

Objectives:

Primary:

* To determine the dose limiting toxicities, toxicity profile, and maximum tolerated dose of CDDO when administered in adult patients with solid tumors and lymphomas.
* To characterize the pharmacokinetics of CDDO.

Secondary:

* To obtain preliminary evidence of anti-tumor activity of CDDO in this population.
* To evaluate the in vivo molecular and biological effects of CDDO by assessing changes in biomarkers of apoptosis and cell cycle arrest.

Eligibility:

* Patients with advance, histological-confirmed malignancies refractory to standard therapy or for which no standard therapy exist.
* Patients should have adequate liver, renal and bone marrow function.

Study Design:

* Accordingly with the accelerated titration design 4B, dose levels will initially be increased at 100% increments, and one new patient per dose level will be treated per 4-week course.
* The accelerated phase ends when one patient experiences DLT during any course of treatment or when two different patients experience grade 2 toxicity during first course of treatment.
* When the first instance of grade 2 toxicity is observed two additional patients must have been treated at that dose, or a higher dose, (during any course) without experiencing moderate or worse toxicity, in order that the accelerated phase continue.
* When the accelerated phase ends, dose-escalation will revert to a more conservative modified Fibonacci scheme with 40% dose-step increments, with at least 3 patients treated per dose level.

DETAILED DESCRIPTION:
Background:

* CDDO is a novel synthetic triterpenoid which is a potent multifunctional molecule. It induces apoptosis in vitro in malignant cells through both intrinsic and extrinsic pathways, and it controls cellular differentiation, apoptosis, and growth inhibition by serving as a ligand for the transcription factor peroxisome proliferator activator receptor-gamma (PPAR gamma).
* Based on in vitro activity, it holds considerable promise as a novel anti-tumor agent against a wide range of malignancies by concurrently targeting multiple pathways leading to oncogenesis.
* In vivo data demonstrates that the drug is well tolerated in dogs, and has anti-tumor effects, dependent upon dose schedule.

Objectives:

Primary:

* To determine the dose limiting toxicities, toxicity profile, and maximum tolerated dose of CDDO when administered in adult patients with solid tumors and lymphomas.
* To characterize the pharmacokinetics of CDDO.

Secondary:

* To obtain preliminary evidence of anti-tumor activity of CDDO in this population.
* To evaluate the in vivo molecular and biological effects of CDDO by assessing changes in biomarkers of apoptosis and cell cycle arrest.

Eligibility:

* Patients with advance, histological-confirmed malignancies refractory to standard therapy or for which no standard therapy exist.
* Patients should have adequate liver, renal and bone marrow function.

Study Design:

* Accordingly with the accelerated titration design 4B, dose levels will initially be increased at 100% increments, and one new patient per dose level will be treated per 4-week course.
* The accelerated phase ends when one patient experiences DLT during any course of treatment or when two different patients experience grade 2 toxicity during first course of treatment.
* When the first instance of grade 2 toxicity is observed two additional patients must have been treated at that dose, or a higher dose, (during any course) without experiencing moderate or worse toxicity, in order that the accelerated phase continue.
* When the accelerated phase ends, dose-escalation will revert to a more conservative modified Fibonacci scheme with 40% dose-step increments, with at least 3 patients treated per dose level.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histologically confirmed (by NIH pathology department) solid tumor malignancy or lymphoma that is metastatic or unresectable and for which there is not therapy with survival benefit and standard curative or palliative measures do not exist.

Patients must have measurable or evaluable disease.

Patients must have recovered less than or equal to grade 1 toxicity levels due to adverse events and/or toxicity of prior chemotherapy or biologic therapy. They must not have had chemotherapy or biologic therapy within 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C, 8 weeks for UCN-01). Patients must be at least 1 month since any prior radiation or major surgery. Patients must be greater than or equal to 2 weeks since any prior participation in a Phase Zero study. Patients on bisphosphonates for any cancer or on androgen deprivation therapy for prostate cancer, however, will not need to discontinue this therapy in order to be eligible.

Age greater than or equal to 18 years.

ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%, see Appendix A).

Life expectancy of greater than 3 months.

Patients must have normal or adequate organ and marrow function as defined below:

* Hb greater than or equal to 10 g/dL
* absolute neutrophil count greater than or equal to 1,500/ L
* platelets greater than or equal to 100,000/ L
* total bilirubin less than or equal to 1.5 normal institutional limits
* AST (SGOT)/ALT (SGPT) less than or equal to 2.5 x institutional upper limit of normal
* creatinine clearance less than 1 x upper limit of normal

OR

-creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.

The effects of CDDO on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation and for 2 months after discontinuation of the study. Women of child bearing potential must have a negative pregnancy test in order to be eligible. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CDDO, breastfeeding should be discontinued if the mother is treated with CDDO.

Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients receiving any other investigational agents.

Patients with known brain metastases are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for at least 6 months after treatment of the brain metastases without steroids or anti-seizure medications. These patients may be enrolled at the discretion of the principal investigator.

History of allergic reactions attributed to other synthetic triperinoids or compounds of similar chemical or biologic composition to CDDO, such as derivative compounds 1-[2-cyano-3-,12- dioxooleana -1,9-dien-28-oyl] imidazole (CDDO-Im), and C-28 methyl ester of 2-cyano-3,12-dioxoolen-1,9-dien-28-oic acid (CDDO-Me).

Patients with clinically significant illnesses which could compromise participation in the study, including, but not limited to: Active or uncontrolled infection, immune deficiencies or confirmed diagnosis of HIV infection, Hepatitis B, Hepatitis C, or uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past six months, uncontrolled cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-05-01; Primary Completion 2008-01-14 (Actual); Study Completion 2008-01-14 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicities, toxicity profile, and maximum tolerated dose of CDDO when administered in adult patients with solid tumors and lymphomas.

SECONDARY OUTCOMES:
To obtain preliminary evidence of anti-tumor activity of CDDO in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ito Y, Pandey P, Sporn MB, Datta R, Kharbanda S, Kufe D. The novel triterpenoid CDDO induces apoptosis and differentiation of human osteosarcoma cells by a caspase-8 dependent mechanism. Mol Pharmacol. 2001 May;59(5):1094-9. doi: 10.1124/mol.59.5.1094. PMID 11306692
- [Background] Lapillonne H, Konopleva M, Tsao T, Gold D, McQueen T, Sutherland RL, Madden T, Andreeff M. Activation of peroxisome proliferator-activated receptor gamma by a novel synthetic triterpenoid 2-cyano-3,12-dioxooleana-1,9-dien-28-oic acid induces growth arrest and apoptosis in breast cancer cells. Cancer Res. 2003 Sep 15;63(18):5926-39. PMID 14522919
- [Background] Ito Y, Pandey P, Place A, Sporn MB, Gribble GW, Honda T, Kharbanda S, Kufe D. The novel triterpenoid 2-cyano-3,12-dioxoolean-1,9-dien-28-oic acid induces apoptosis of human myeloid leukemia cells by a caspase-8-dependent mechanism. Cell Growth Differ. 2000 May;11(5):261-7. PMID 10845427